CLINICAL TRIAL: NCT03885986
Title: Ultrasound Evaluation of Cysts and "Cyst-like" Lesions in and Around the Knee:In Comparison to Magnetic Resonance Imaging
Brief Title: Ultrasound Evaluation of Cystic Lesions in the Knee:In Comparison to Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Bahaa Boshra, Principal Investigator, Assiut University
Other Study IDs: US,MRI of knee cysts
Record Dates: First submitted 2019-03-18; First posted 2019-03-22 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Knee Cyst Popliteal (___Cm)
MeSH Terms: conditions — Popliteal Cyst | interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Ultrasound — role of ultrasound in comparison to magnetic resonance imaging in diagnosis of benign cystic lesions of knee
  Other Names: magnetic resonance imaging

SUMMARY:
Benign cysts and cystic-appearing lesions in and around the knee are common and differentiation between them through the history, symptoms and clinical examination is difficult due to the presence of common findings such as pain, edema, and palpable mass. The clinical presentation depends on the location, size of the lesion and its relation with the surrounding structures.

DETAILED DESCRIPTION:
The Benign knee cysts can be subdivided into four major categories as following:1- synovial cysts, 2- popliteal (Baker's) cyst, 3- ganglion cysts, 4- meniscal cysts. Whereas, The "cyst-like" lesions can be sub-classified into the following:1- normal knee bursae, 2- normal knee recesses, 3- miscellaneous cyst-like lesions as aneurysms, hematomas, seromas and abscess.

Many of these lesions have fairly characteristic locations and imaging features. Knowledge of these variants and lesions is essential for accurate diagnosis and to avoid mistaking them for aggressive soft tissue lesions, including sarcomas. Ultrasonography and magnetic resonance imaging are the most useful imaging modalities in evaluating these Benign cystic lesions. Ultrasonography can distinguish cysts from solid lesions and assess the degree of vascularity within the lesion. Magnetic resonance imaging can help to delineate the location of the lesion in relation to anatomic structures and also determine if the lesion is cystic or solid when contrast is administered.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosed cystic lesions in and around the knee.

Exclusion Criteria:

1. arthroscopy or surgical intervention to the knee joint.
2. fracture repaired by metal plates or screws.
3. claustrophobia.
4. contraindications to MRI as patients with implanted pacemaker or defibrillator, ferromagnetic aneurysm clips and metallic foreign body at the knee joint.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients in different age groups referred to Radiology department at Assiut University Hospital with clinically suspected benign cystic lesions in and around the knee.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Role of ultrasound and magnetic resonance imaging in diagnosis of Benign knee cysts | within 3 hours
  Results of ultrasound in comparison to results of magnetic resonance imaging in diagnosis of Benign knee cysts.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perdikakis E, Skiadas V. MRI characteristics of cysts and "cyst-like" lesions in and around the knee: what the radiologist needs to know. Insights Imaging. 2013 Jun;4(3):257-72. doi: 10.1007/s13244-013-0240-1. Epub 2013 Mar 12. PMID 23479129
- [Background] Telischak NA, Wu JS, Eisenberg RL. Cysts and cystic-appearing lesions of the knee: A pictorial essay. Indian J Radiol Imaging. 2014 Apr;24(2):182-91. doi: 10.4103/0971-3026.134413. PMID 25024531
- [Background] Wu JS, Hochman MG. Soft-tissue tumors and tumorlike lesions: a systematic imaging approach. Radiology. 2009 Nov;253(2):297-316. doi: 10.1148/radiol.2532081199. PMID 19864525
- [Background] Bermejo A, De Bustamante TD, Martinez A, Carrera R, Zabia E, Manjon P. MR imaging in the evaluation of cystic-appearing soft-tissue masses of the extremities. Radiographics. 2013 May;33(3):833-55. doi: 10.1148/rg.333115062. PMID 23674777
- [Background] Steinbach LS, Stevens KJ. Imaging of cysts and bursae about the knee. Radiol Clin North Am. 2013 May;51(3):433-54. doi: 10.1016/j.rcl.2012.10.005. Epub 2013 Jan 12. PMID 23622093
- [Background] Alessi S, Depaoli R, Canepari M, Bartolucci F, Zacchino M, Draghi F. Baker's cyst in pediatric patients: Ultrasonographic characteristics. J Ultrasound. 2012 Feb;15(1):76-81. doi: 10.1016/j.jus.2011.06.007. Epub 2011 Jul 1. PMID 23396996